CLINICAL TRIAL: NCT03030326
Title: Biofeedback for Asthma Comorbid With Anxiety or Depression
Acronym: ASANX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding to hire staff, could not find student to do project
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Paul Lehrer, Ph.D., Professor of Psychiatry, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20160001007
Record Dates: First submitted 2016-09-15; First posted 2017-01-25 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: ASTHMA; ANXIETY
MeSH Terms: conditions — Asthma; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart rate variability biofeedback (Experimental): This group will receive treatment in the first three months of the study and will be observed during the second three months
  Interventions: Behavioral: heart rate variability biofeedback
- Observation first (No Intervention): This group will be observed during the first three months and given biofeedback during the second three months

INTERVENTIONS:
Behavioral: heart rate variability biofeedback — Patients learn to increase heart rate variability by breathing at the resonance frequency of the cardiovascular system, at approximately 6 breaths/min, varying among people.
  Arms: Heart rate variability biofeedback

SUMMARY:
Twenty patients with a history of treatment, within the past year, of both asthma and either depression or an anxiety disorder will be recruited for this study. Patients will be recruited from their doctors and from advertisements. The investigators will randomly assign patients to two groups, using a crossover design. One group will first receive three months with four biweekly sessions of heart rate variability biofeedback treatment, and then will be followed for three months with a daily symptom diary. The other group will first be followed for three months, and then given the three months of treatment. In both treatment and following procedures, patients will receive psychophysiological testing sessions at the beginning and end of the three month period. The investigators will assess symptoms of asthma, anxiety, and depression as well as pulmonary function and will measure heart rate (from electrodes on the wrists), respiration (through a belt around the waist), end tidal carbon dioxide (through a cannula in the nose).

DETAILED DESCRIPTION:
Introduction

Previous published research from our laboratory has demonstrated a clinically significant effect for heart rate variability biofeedback on asthma clinical condition. In an NIH-supported trial just completed, however, the investigators found that, among unmedicated patients with mild or moderate asthma, the effects were no greater than for most placebos found in the literature. Significant effects were found in reducing anxiety and depression, even among a population that was selected neither for clinical anxiety or depression.

There is considerable evidence from the literature that negative affect is common in asthma, and that it may interact with asthma. Anxiety is often accompanied by hyperventilation, as is asthma, and hyperventilation can exacerbate asthma, by increasing exposure to in air that is colder drier than the lung (body temperature at 100% humidity). Indeed some of the asthma symptoms affecting quality of life are associated with hyperventilation, which may partially be stimulated by anxiety, and partially by increased airway resistance, which increases respiratory drive. Thus asthma processes can increase anxiety (through symptoms associated with hyperventilation), just as anxiety can exacerbate asthma (through hyperventilation). Additionally, autonomic hyperreactivity, which is common in anxiety, may produce parasympathetic hyperreactivity that may cause bronchoconstriction. There is considerable evidence that heart rate variability (HRVB) biofeedback ameliorates anxiety, just as it does asthma, so the combined effect may prove particularly beneficial to people with the comorbid condition. The investigators therefore propose a pilot study to test the effect of HRVB on an asthma population that is clinically anxious.

Another consistent effect of HRVB is on ameliorating depression. There is a good physiological rationale for using HRVB to treat negative affect and depression, stemming from anatomical evidence for connections between the site of HRVB effects on the baroreflex (mediated through nucleus tractus solitarius) and brain centers involved in negative emotion, particularly the insula and amygdala. Depression also is highly prevalent among asthma patients, and depressed patients often have poor health care behavior, and this may worsen asthma condition. Depressive symptoms also are associated with bronchoconstriction in asthma. Anxiety and depression are frequently comorbid, with some overlapping symptoms, so many anxiety patients will be expected to also show signs of clinical depression.

Also, it is possible that HRVB may improve by making asthma medication more available to the lungs, through deep breathing. Therefore asthma medication will not be restricted in this study, but medication intake will be monitored as one outcome measure. Similarly medication for anxiety or depression also will not be controlled, but daily intake and changes in medications will be monitored. Additionally patients with all levels of asthma severity will be studied, as long as they continue to be symptomatic. It is possible that, in a previous study, restricting inclusion to patients only with very mild asthma may have contributed to a floor effect that obscured biofeedback effects.

In this study the investigators will use the same HRVB protocol as used in previous studies. The control group will be a waiting list control, who will be given a post-assessment at three months, and then given the treatment protocol, in a crossover design.

Study Duration: 6 months

Subject Recruitment and Selection:

Twenty patients will be recruited for this study, 10 for the treatment group and 10 for the control group.

Subjects will be recruited from media advertisements, physician referrals, and from letters (approved by the Institutional Review Board) sent by physicians to their asthma patients inviting them to participate in the study. At the physicians' request, study personnel may assist the office in preparing mailings. The investigators also will work with a large behavioral healthcare organization, University Behavioral Healthcare (UBHC), which also provides primary care to patients treated there. UBHC will provide a list of patients with diagnoses including asthma and one of the anxiety disorders. The investigators will contact the patient's physician or therapist, and ask the provider to give a recruitment brochure to the patient, inviting the patient to call the study.

Methods

The study will take place over a course of six months.

Screening and run-in. At the first session, patients will first be consented. Then they will be given an interview to determine medical and psychiatric history, and will be given the Asthma Control Test and the Beck Anxiety Inventory. They also will be given a peak flow meter, trained to take a reliable measure with it, and instructed in completing the daily diary. Patients who are unable to follow these procedures by the following session (about 1-2 weeks later, the first psychophysiological test session, as described below) will be screened out. Patients will be administered the Asthma Quality of Life questionnaire for standardized situations, Asthma Control Test, the Beck Depression Inventory and the Beck Anxiety Inventory. The Marlowe-Crowne Social Desirability Scale also will be administered in the pretest session, as this test is known to predict the correlation between symptoms self report and psychophysiological indicators, as well as stress-related asthma symptomatology.

First three month treatment phase: Treatment and control procedures will take place in the first three months, The three months of treatment will consist of 5 biweekly treatment sessions, and 2 measurement sessions (with a third session for patients in the control group after they receive treatment). In the control condition, patients will be asked to send daily questionnaires (and be given reminder calls) every two weeks). They will be provided with stamped addressed envelopes. The treatment sessions will be an hour long each and the measurement sessions will be 2 hours long.

Second three-month treatment phase: Following the post-test psychophysiological test session, subjects in the control condition will be given three months of treatment, as above, and patients initially assigned to the Treatment group will receive the same procedure as control group subjects in the initial phase.

Home practice: Subjects will be asked to do paced breathing at their resonance frequency (approximately 6 breaths/min) for 20 min twice daily after the first session of treatment. Subjects who find this procedure difficult will be lent a biofeedback machine for home practice.

Psychophysiological testing sessions

Psychophysiological testing sessions will take place before the first treatment session (or waiting list period), and after the last treatment session (or waiting list period) in both phases of the study. Thus three testing sessions will be given.

Questionnaires: In the second and third testing sessions, the same questionnaires given at the screening session will be readministered.

A pulmonary function test will be performed using standard spirometry (Three forced expiratory maneuvers from maximal vital capacity). Sensors will then be affixed to measure heart rate (from the wrists), respiration (a strain gauge around the waist), finger pulse volume (from a plethysmograph attached to the middle finger of the nondominant hand), and palmar skin conductance (from electrodes pasted to the forefinger and thenar eminence of the nondominant hand). Exhaled carbon dioxide will be collected from a nasal cannula to measure hyperventilation symptoms, which are targeted by HRVB, and which are common in asthma.

After sensors are attached, 5-min baseline period will take place in which patients will do a 'plain vanilla task' (looking at a series of colored rectangles, counting the number of a particular color), followed by 5 minutes of HRV biofeedback or uninstructed relaxation (for the control group), followed by another baseline. After each 5-min period, three minutes of testing will be done using a forced oscillation pneumograph, followed by spirometry (the standard 3-puff procedure). This instrument involves playing sound waves into the mouth, and measuring sounds bounced back from the lung.

Because the canulas are sometimes mildly uncomfortable, the 5-min baseline and biofeedback (or relaxation) periods will be given twice, once with the measure of end tidal carbon dioxide (CO2) and once without.

Testing sessions will be performed after a 6-hour albuterol withhold. If a patient experiences an exacerbation of asthma symptoms, the patient will be instructed to take medication as usual, and the session will be rescheduled.

Pulmonary function measures (impulse oscillometry and spirometry) will be taken using a Jaeger 'IOS (Impulse Oscillometry System) Masterscreen' unit after each 5-min assessment period. Other psychophysiological measures will be taken using a J&J Engineering C2+, which will output electrocardiogram (EKG) data at 1000 samples/sec for later analysis using a program called 'WinCPRS'.

Daily measures

Patients will be asked to provide a daily symptom diary and twice daily peak flow readings (morning upon arising and evening prior to retiring)

Randomization

A stratified randomization protocol will be used, with three criteria: gender, age (older or younger than 40, the age where HRV tends to abruptly decrease), and asthma control (percent expected on the basis of normative data of the amount of air exhaled in the first second of a forced expiratory maneuver from maximal vital capacity (FEV1).

Statistical treatment

A mixed models repeated measures analysis will be done on all measures with Treatment as a between-groups measure and Session (and Task for physiological measures after the three tasks in the physiological testing sessions).

ELIGIBILITY:
Inclusion Criteria:

* Asthma: A diagnosis of asthma within the past year, and any of the following: history of a previous positive methacholine challenge test, or history of a positive response to albuterol and/or inhaled or oral steroid medication. We only will accept patients whose asthma is not under complete control, so an additional criterion will be an Asthma Control Test score of < 19.
* Age: 18-75.
* Anxiety: A Beck Anxiety Scale score ≥ 10 (mild anxiety) and a history of medical or psychological treatment of anxiety within the past year.

Exclusion Criteria:

* Comorbid disease. A diagnosed lung disease other than asthma, a cardiac rhythm disturbance (e.g., frequent preventricular or preatrial contractions, mitral valve prolapse, active psychosis, taking antipsychotic medications, presence of other serious or life threatening disease (e.g., cancer, or serious renal, hepatic, cardiac, immunodeficiency, neurological, or other disease), epileptic seizure within the past year
* Asthma Severity: Hospitalization for asthma within the past year.
* Linguistic and intellectual competence. Inability to understand English, illiteracy, or mental incapacity, understand informed consent procedures, or complete questionnaires or follow procedures.
* Smoking: Patients must be non-smokers for at least the past year and have less than a 15 pack-year smoking history.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-10 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change in asthma control test | From pretest to 3 and 6 months (after the treatment or waiting list phase, respectively, repeated at crossover)
  paper and pencil scale of asthma symptoms. This study uses a crossover design. the first post-test is at 3 months. Then the conditions are switched, such that the experimental group gets the control condition and the control group gets the experimental condition. The measure will then be taken 3 months later, i.e. at the 6 month period.
change in Beck Anxiety Inventory | Pretest to 3 and 6 months (after the treatment or waiting list phase, respectively, repeated at crossover)
  paper and pencil scale of anxiety symptoms. This study uses a crossover design. the first post-test is at 3 months. Then the conditions are switched, such that the experimental group gets the control condition and the control group gets the experimental condition. The measure will then be taken 3 months later, i.e. at the 6 month period.
change in Beck Depression Inventory | Pretest to 3 and 6 months (after the treatment or waiting list phase, respectively, repeated at crossover)
  paper and pencil scale of depression symptoms. This study uses a crossover design. the first post-test is at 3 months. Then the conditions are switched, such that the experimental group gets the control condition and the control group gets the experimental condition. The measure will then be taken 3 months later, i.e. at the 6 month period.

SECONDARY OUTCOMES:
change in forced oscillation pneumography (resistance to 5 - 35 Hz sound stimulation | Pretest to approximately 3 and 6 months (after the treatment or waiting list phase, respectively, repeated at crossover)
  Patients will be tested for three minutes on a forced oscillation pneumograph after a 5-min rest period and after a 5-min biofeedback period (or self-relaxation, for patient who have not been trained yet)
Daily symptoms throughout participation in the study ( changes over 6 months) | Daily from pretest to last session, approximately 6 months
  Paper and pencil scale of asthma symptoms
Home peak flow readings taken twice daily between 1st and last sessions (changes over 6 months) each subject | At pretest and daily for 6 months of participation in the study
  Patients blow into a peak flow meter as hard and fast as possible, three times for each measure, once just after arising in the morning and one just before retiring in the evening
Spirometry, where we measure FEV1 (changes over 6 months the volume of air exhaled during the first second of a forced expiratory maneuver from maximal vital capacity) | At pretest and at 3 and 6 months (after the treatment or waiting list phase, respectively, repeated at crossover)
  Patient blows into a peak flow meter as hard and fast as possible from the deepest breath possible three times at each assessment. This study uses a crossover design. the first post-test is at 3 months. Then the conditions are switched, such that the experimental group gets the control condition and the control group gets the experimental condition. The measure will then be taken 3 months later, i.e. at the 6 month period.
Low frequency heart rate variability | At pretest and 3 and 6 months (changes within session and over time) after the treatment or waiting list phase, respectively, repeated at crossover)
  Spectral amplitude of interbeat cardiac intervals between 0.05 - 0.15 Hz recorded from the R-spike of the electrocardiogram. This study uses a crossover design. the first post-test is at 3 months. Then the conditions are switched, such that the experimental group gets the control condition and the control group gets the experimental condition. The measure will then be taken 3 months later, i.e. at the 6 month period.
End tidal carbon dioxide (CO2) | Changes within session and over time, taken at pretest and 3 and 6 months (after the treatment or waiting list phase, respectively, repeated at crossover)
  Taken on a capnometer through a nasal canula immediately after each 5 -min task (baseline or biofeedback). This study uses a crossover design. the first post-test is at 3 months. Then the conditions are switched, such that the experimental group gets the control condition and the control group gets the experimental condition. The measure will then be taken 3 months later, i.e. at the 6 month period.
Marlowe Crowne Social Desirability Scale | Given only at the pretest session
  This is a suppressor variable not an outcome variable. It is given only once and used as a covariate for other measures

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lehrer, PhD, Study Director — Rutgers Health Sciences IRB - New Brunswick/ Piscataway campus

IPD SHARING:
Plan to Share IPD: Undecided
We hope to publish data.